CLINICAL TRIAL: NCT06002997
Title: Periodontal Status and Pregnancy or Delivery Complications in Type 1 Diabetes Mellitus Pregnant Women: a Case-control Study From Slovenia
Brief Title: Periodontal Status and Pregnancy or Delivery Complications in Type 1 Diabetes Mellitus Pregnant Women
Status: Completed | Type: Observational
Sponsor: University of Ljubljana (Other)
Collaborators: University Medical Centre Ljubljana (Other)
Responsible Party: Sponsor
Other Study IDs: Pregnancy, DM, Periodontitis
Record Dates: First submitted 2023-05-08; First posted 2023-08-21 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Periodontal Diseases; Periodontitis; Pregnancy Complications; Pregnancy in Diabetic; Diabetes Mellitus, Type 1; Delivery Complication
Keywords: Periodontal disease; Type 1 Diabetes Mellitus; C-section; Gestational Week of Birth
MeSH Terms: conditions — Periodontal Diseases; Periodontitis; Pregnancy Complications; Pregnancy in Diabetics; Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Group: Healthy pregnant women
  Interventions: Other: Pregnancy and/or delivery complications; Other: Periodontal disease
- Case Group: Pregnant women with Diabetes Mellitus Type 1
  Interventions: Other: Pregnancy and/or delivery complications; Other: Periodontal disease

INTERVENTIONS:
Other: Pregnancy and/or delivery complications — Analysis of post-delivery reports for pregnancy and/or delivery complications.
Other: Periodontal disease — Measuring clinical periodontal parameters for assessing presence of periodontal disease.

SUMMARY:
The results of contemporary studies suggest an association between inflammatory periodontal disease and pregnancy and delivery complications. The aim of this study was to assess the association between periodontal disease, clinical periodontal parameters and pregnancy or delivery complications in type 1 diabetes mellitus and non-diabetic pregnant women.

DETAILED DESCRIPTION:
The results of contemporary studies suggest an association between inflammatory periodontal disease and pregnancy and delivery complications. The aim of this study was to assess the association between periodontal disease, clinical periodontal parameters and pregnancy or delivery complications in type 1 diabetes mellitus and non-diabetic pregnant women. Methods: 15 type 1 diabetes mellitus and 15 non-diabetic primiparous women were enrolled in the prospective "case-control" study. Investigators compared periodontal status, levels of glycosylated haemoglobin (HbA1c), high sensitivity C-Reactive Protein (hs-CRP), gestational week of birth, birth weight of a newborn and pregnancy or delivery complications (C-section, pre-eclampsia) between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Pregnant Women
* Pregnant Women with Diabetes Mellitus type 1
* Healthy Pregnant Women with signs of Periodontal Disease
* Pregnant Women with Diabetes Mellitus type 1 and signs of Periodontal disease

Exclusion Criteria:

* Smokers
* Former smokers who had stopped smoking less than five years before participation
* Pregnant women with other systemic diseases

Max Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Pregnant women included in study entitled: Periodontal status of type 1 diabetes mellitus and healthy pregnant women: a case-control study from Slovenia
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-05-03 (Actual); Primary Completion 2014-12-01 (Actual); Study Completion 2014-12-01 (Actual)

PRIMARY OUTCOMES:
Number of Delivery and/or Pregnancy complications | Day of delivery
  Yes/No
Number of C-section | Day of delivery
  Yes/No
Number of pregnant women with Pre-eclampsia | Between 28th and 34th week of gestation
  Yes/No
Number of Pre-term births GWOB (Gestational week of birth) ≤ 37th week | Day of delivery
  Yes/No
GWOB - Gestational week of birth | Day of delivery
  Week number
number of Births with weight ≤ 2500 g | Day of delivery
  Yes/No
Birth weight | Day of delivery
  Weight in kg
Number of pregnant women with Periodontal disease | Between 28th and 34th week of gestation
  Yes/No

SECONDARY OUTCOMES:
Age | Between 28th and 34th week of gestation
  Age
BMI (Body mass index) | Between 28th and 34th week of gestation
  Body mass index - measure of body fat based on height and weight (BMI = Weight (kg) / Height (m)²)
PPD (Probing pocket depth) | Between 28th and 34th week of gestation
  Probing pocket depth (measured on 6 sites around teeth, unit: mm)
CAL (Clinical attachment loss) | Between 28th and 34th week of gestation
  Clinical attachment loss (measured on 6 sites around teeth, unit: mm) - This is the measurement of the position of the soft tissue attachment in relation to the cemento-enamel junction (CEJ). Two measurements are used to calculate the CAL: the probing depth and the distance from the gingival margin to the CEJ.
percantage of sites with BOP (Bleeding on probing) | Between 28th and 34th week of gestation
  Bleeding on probing, Yes/No after probing pocket depth measurement 6 sites around each tooth. Unit: %
TPIB (Total periodontal inflammatory burden) | Between 28th and 34th week of gestation
  Total periodontal inflammatory burden - measures of average teeth neck circumferences by tooth type, probing depth (PD) and bleeding on probing (BOP). The subgingival area for each tooth was calculated by multiplying 1/6th of the average cervical circumference of the tooth with each of the six measurements of probing depth. The sum of subgingival areas of all present teeth in a subject represented the total subgingival area of an individual.
TBPW area (Total bleeding periodontal wound) | Between 28th and 34th week of gestation
  Total bleeding periodontal wound - measures of average teeth neck circumferences by tooth type, probing depth (PD) and bleeding on probing (BOP). The subgingival area for each tooth was calculated by multiplying 1/6th of the average cervical circumference of the tooth with each of the six measurements of probing depth. The sum of subgingival bleeding areas of all present teeth in a subject represented the total subgingival area of an individual.
Percantage of HbA1C (Glycosylated haemoglobin) | Between 28th and 34th week of gestation
  Glycosylated haemoglobin, Unit: %

CONTACTS AND LOCATIONS:
Overall Officials: Rok Schara, DMD, PhD, Study Director — Assistant Professor

IPD SHARING:
Plan to Share IPD: No
All Research data will be available or shared on individual request. Example: conducting Meta-Analysis.

REFERENCES:
- [Background] Bassani DG, Olinto MT, Kreiger N. Periodontal disease and perinatal outcomes: a case-control study. J Clin Periodontol. 2007 Jan;34(1):31-9. doi: 10.1111/j.1600-051X.2006.01012.x. Epub 2006 Nov 20. PMID 17116160
- [Background] Bosnjak A, Relja T, Vucicevic-Boras V, Plasaj H, Plancak D. Pre-term delivery and periodontal disease: a case-control study from Croatia. J Clin Periodontol. 2006 Oct;33(10):710-6. doi: 10.1111/j.1600-051X.2006.00977.x. Epub 2006 Aug 3. PMID 16889630
- [Background] Sacco G, Carmagnola D, Abati S, Luglio PF, Ottolenghi L, Villa A, Maida C, Campus G. Periodontal disease and preterm birth relationship: a review of the literature. Minerva Stomatol. 2008 May;57(5):233-46, 246-50. English, Italian. PMID 18496486
- [Background] Champagne CM, Madianos PN, Lieff S, Murtha AP, Beck JD, Offenbacher S. Periodontal medicine: emerging concepts in pregnancy outcomes. J Int Acad Periodontol. 2000 Jan;2(1):9-13. PMID 12666980
- [Background] Ide M, Papapanou PN. Epidemiology of association between maternal periodontal disease and adverse pregnancy outcomes--systematic review. J Periodontol. 2013 Apr;84(4 Suppl):S181-94. doi: 10.1902/jop.2013.134009. PMID 23631578
- [Background] Ruma M, Boggess K, Moss K, Jared H, Murtha A, Beck J, Offenbacher S. Maternal periodontal disease, systemic inflammation, and risk for preeclampsia. Am J Obstet Gynecol. 2008 Apr;198(4):389.e1-5. doi: 10.1016/j.ajog.2007.12.002. Epub 2008 Mar 4. PMID 18295179